CLINICAL TRIAL: NCT06282783
Title: A Phase I/II Clinical Trial Investigating the Effect of Topiramate on the Reactivation of the HIV-1 Reservoir in People Living With HIV on Antiretroviral Therapy
Brief Title: Studying Topiramate for Re-Activating the HIV-1 Reservoir
Acronym: STAR
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Casper Rokx, Associate Professor, Erasmus Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-511532-27-00
Record Dates: First submitted 2024-02-12; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: HIV-1-infection; Hiv; HIV Infections; HIV I Infection
Keywords: HIV Cure; Shock and Kill; Topiramate; Latency Reversing Agents; Latency Reversal
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections; Shock | interventions — Topiramate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Men (Experimental): Sex assigned at birth, male Single dose of 400mg topiramate
  Interventions: Drug: Topiramate
- Women (Experimental): Sex assigned at birth, female Single dose of 400mg topiramate
  Interventions: Drug: Topiramate

INTERVENTIONS:
Drug: Topiramate — Single dose of 400mg

SUMMARY:
Even with current HIV treatments, HIV is still a lifelong disease because it hides in some long-lasting cells in the body. One of the strategies to find a cure for HIV works by finding the virus in these cells, making it visible, and then getting rid of it. This is called the 'shock and kill' approach.

So far, the drugs tested can find the virus, but they don't get rid of it completely. That's why there need to be new drugs that can do this more effectively. The Erasmus MC HIV Eradication Group (EHEG) has been testing new drugs in the lab and found a drug called topiramate can wake up the virus without harming the cells. The aim of this study is to test topiramate in people living with HIV.

Most of the people that participate in HIV cure studies are men, even though most people living with HIV around the world are women. Previous research has shown that men and women might respond differently to these treatments. So, in this study, topiramate will be investigated in both men and women. This could help us find a cure that works for everyone.

DETAILED DESCRIPTION:
Despite antiretroviral therapy (ART), an infection with the human immunodeficiency virus 1 (HIV-1) is still a lifelong disease because of the latent HIV reservoir. This reservoir consists of a pool of long-lived cells harbouring an integrated copy of the HIV provirus in its genome. One approach to curing HIV centres on reversing viral latency, combined with the subsequent elimination of the virus from this reservoir specifically, all while safeguarding other cells through the use of ART. This approach is colloquially known as 'shock and kill'. The limited number of latency reversing agents (LRAs) that have been studied were effective at reactivating the latent reservoir, but do not result in significant reservoir reduction (Debrabander, 2023). Investigating novel LRAs is, therefore, necessary to identify more potent ways of HIV reactivation, with the ultimate goal of reservoir depletion i.e. a functional HIV cure. The Erasmus MC HIV Eradication group has set up a translational trial platform, where successfully study the effects of novel LRAs from bench to bedside. One example is the discovery of small molecule inhibitors of BAF, which reverse HIV-1 latency, to a clinical trial investigating pyrimethamine in people living with HIV (PLWH) (Stoszko, 2016; Prins, 2023). A new promising drug target that was identified in EHEG is the glutamate receptor, ionotropic kainate 5 (GRIK5); a host factor involved in HIV latency (Roling, 2021). The registered drug topiramate was identified as a potential GRIK5 inhibitor. Further ex vivo testing confirmed HIV latency reversal of topiramate at therapeutic levels without inducing cytotoxic effects. This opens new opportunities for HIV cure research. A further knowledge gap to be explored is the influence of sex in HIV latency reversal. Typically, either by design or recruitment, male participants have been vastly overrepresented in HIV cure research (Barr, 2020). This is despite previous research showing significant difference in HIV latency reversal in women (Rao, 2022), and the importance of sex in pharmacodynamics being increasingly recognised (Gandhi, 2004; Mauvais-Jarvis, 2021). As the majority of PLWH worldwide are women and their numbers are expected to grow, studies on any potential cure strategy that provide an evidence base for their use in women increase clinical impact (UNAIDS, 2023). Therefore, the aim of this study is to examine the effect and safety of topiramate as an LRA in both men and women.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV-1, subtype B or C
* Aged 18 or over
* On ART for a minimum of 2 consecutive years and a maximum of 12 consecutive years
* HIV-1 RNA plasma level <30 copies/mL for at least two consecutive measurements prior to inclusion (viral blips with a detectable HIVRNA 30-200 c/mL preceded and followed by HIV-RNA <30 are allowed)
* CD4+ T cell count ≥200 cells/mm^3 at screening
* Able to understand the information and give informed consent

Exclusion Criteria:

* Any major acute medical condition requiring hospitalisation within the past 4 weeks.
* Presence of an active opportunistic infection that defines Acquired Immunodeficiency Syndrome (AIDS).
* Any medical condition deemed by the investigator to hinder compliance with the study treatment.
* The following laboratory values at the screening phase (available before baseline (T0)): hepatic transaminases (AST or ALT) ≥3 times the upper limit of normal (ULN), serum total bilirubin ≥3 times the ULN, estimated glomerular filtration rate (eGFR) ≤60 mL/min based on CKD-EPI, haemoglobin <6.5 mmol/L (males) or <6.0 mmol/L (females), leucocytes <2.5 x10^9/L, absolute neutrophil count <1000 cells/mm^3, thrombocytes <100 x10^9/L
* Active malignancy during the past year except for basal carcinoma of the skin, stage 0 cervical carcinoma, Kaposi Sarcoma treated with ART alone, or other indolent malignancies.
* Participants who are unwilling or unable to use barrier contraception during sexual intercourse during the study.
* History of suicide or suicidal ideation.
* History of ophthalmological medical problems leading to glaucoma or visual field disturbances (e.g. macula oedema). Refraction abnormalities that can be corrected by lenses are acceptable.
* History of any medical condition with a causal relationship with hyperammonemia.
* Participants using phenytoin, carbamazepine, digoxin, lithium, or valproic acid throughout the trial period.
* Any concurrent medicine use associated with hyperammonemia (e.g. valproic acid).
* Participants with active substance abuse.
* Participants who have registered allergies to the investigational medical product.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Effect of topiramate as measured by cell-associated HIV RNA | 24 hours
  To assess the effect of topiramate on HIV reactivation in people living with HIV on ART
Number of treatment-related adverse events as assessed by CTCAE v4.0 | 7 days
  To evaluate the clinical safety and tolerability of topiramate

SECONDARY OUTCOMES:
Influence of sex on the primary outcome measures | 24 hours
  To evaluate the influence of sex on reactivation potential as measured by cell-associated HIV RNA, and safety and tolerability of topiramate as assessed by CTCAE v4.0
The effect of topiramate on the size of the HIV reservoir measured by relevant assays | 24 hours
  To assess the effect of topiramate on the size of the HIV reservoir

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus Medical Centre, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
The data will be stored in accordance with the FAIR use principle for potential future studies. If external researchers express interest in this dataset, they are encouraged to reach out to the lead investigator. Provided that sufficient privacy measures are in place, the data may be disseminated under a newly established Data Sharing Agreement.